CLINICAL TRIAL: NCT04266002
Title: Prospective Study in HIV-1 Infected Adult Subjects With HIV-associated Neurocognitive Disorders Despite Effective Antiretroviral Therapy in Plasma, After a Change in HIV Treatment With an Increased of CHARTER Score ≥ 3 (Total Score ≥ 9)
Brief Title: HIV-1 Infected Adult Subjects With HIV-associated Neurocognitive Disorders Despite Effective Antiretroviral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Franco-Britannique-Fondation Cognacq-Jay (Other)
Collaborators: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Gilles Force, MD, Study promotor, Hôpital Franco-Britannique-Fondation Cognacq-Jay
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHFB001
Record Dates: First submitted 2020-01-24; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: HIV-1-infection; HIV Associated Neurocognitive Disorder
Keywords: CNS Penetration Effectiveness; Global Deficit Score; Cytokines; CSF Inflammation

STUDY DESIGN:
Intervention Model Description: Prospective Pilot study, open-label, multicenter in the Ile-de-France
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIV-1 infected adult associated neurocognitiv (Other): HIV-1 infected adult subjects with HIV-associated neurocognitive disorders despite effective antiretroviral therapy in plasma for more than one year, analyzing the evolution of cognitive disorders with Global Deficit Score and HAND classification, and markers of macrophagic inflammation in blood and cerebrospinal fluid, after a change in HIV treatment with an increased of the new scale CHARTER score ≥ 3 (total treatment score to be ≥ 9)
  Interventions: Other: Validation of Charter score for the CNS diffusion of antiretroviral drugs

INTERVENTIONS:
Other: Validation of Charter score for the CNS diffusion of antiretroviral drugs — IHFB001 (Neuroplustrois) is a pilot study, phase IV, open-label, multicenter in Ile-de-France region, trying to demonstrate the improvement of cognitive change after treatment characterized by its better diffusion in the central nervous system. The characteristics of the change in treatment are (Cn - Ci) ≥ 3 and Cn ≥ 9, where Cn is the Charter score of the new treatment and Ci the Charter score of the initial treatment.

SUMMARY:
Prospective study in HIV-1 infected adult subjects with HIV-associated neurocognitive disorders despite effective antiretroviral therapy in plasma for more than one year, analyzing the evolution of cognitive disorders and markers of macrophagic inflammation in blood and cerebrospinal fluid, after a change in HIV treatment with an increased of the new scale CHARTER score ≥ 3 (total treatment score to be ≥ 9)

DETAILED DESCRIPTION:
Neurocognitive disorders are measured using Frascati 3-stage classification and Global Deficit Score, after the following 10 standardized battery test: Grooved Pegboard for dominant and non-dominant hand, Grefex Verbal Fluency, California Verbal Learning Test (CVLT), Digit Span Wechsler Adult Intelligence Scale III, modified Paced Auditory Serial Addition Test (60 items), WAIS III Digit Symbol Test, Trail Making Test A&B, recall of CVLT and Wisconsin Card Sorting Test; and after the Beck Depression Inventory II (BDI), Inventory of Activity Daily Living part II (IADL) and 10-items Cognitive Complaint Questionnaire (CCQ). The global CNS Penetration Effectiveness (CPE) score of ARV treatment are the sum of the scores of each ARV the patient received, according to the last published scoring. For each drug class, we considered treatment intensification only for drugs with CPE score reaching at least 3 (no intensification if switch in same drug class with same CPE score). CPE score was corrected by drugs resistance status, using cumulative genotype interpreted with the 2012 ANRS algorithm (www.hivfrenchresistance.org; v.2012) at inclusion (CPE=0 if resistance).

ELIGIBILITY:
Inclusion Criteria:

1. Subject (male or female) with HIV-1 infection
2. Subject is ≥ 18 years of age
3. Subject with a plasma viral load (HIV-1 RNA) undetectable for at least one year or with minimal replication <500 copies/ml for at least one year at the inclusion date
4. Patient with HIV-associated neurocognitive disorders : at least two ability domains, documented by performance of at least 1.0 standard deviation below the mean for age-education appropriate norms on standardized neuropsychological tests
5. Patient is willing and able to understand and provide written informed consent prior to participation in this study

Exclusion Criteria:

1. Subject with HIV-2 infection
2. Subject with plasma viral load (HIV-1 RNA)> 500 copies/ml in the past year
3. Subject with acquired impairment in cognitive functioning involving only one ability domain, or involving at least two ability domains but with performance better than 1.0 standard deviation below the mean (no evidence of potential cognitive impairment)
4. Subject unable, according to the investigator, to meet the study requirements, including patients unable to perform cognitive tests
5. Subject with acute intercurrent disease
6. Patient with positive serology for HCV or HBsAg positive
7. Subject with cognitive impairment related to another cause than HIV: other CNS infection, CNS neoplasm, cerebrovascular disease, preexisting neurologic disease or metabolic disorders, severe substance abuse, or systemic disease.
8. Subject with a brain MRI or CSF analysis results that suggest another pathology than HIV associated neurocognitive disorder
9. Subject requires treatment with immunomodulating agents (or may require such treatment during the two years monitoring) such as systemic corticosteroïds, interferons, interleukins, growth factor GM- CSF, or other targeted therapy that may interfere with macrophage markers of the study
10. Subject requires treatment with radiation therapy or cytotoxic chemotherapeutic agents
11. Subject at which the initial lumbar punction can't be achieved
12. Subject ≥65 years at the inclusion date, age with high risk of atherosclerotic disease
13. Subject with significant depression : with a score ≥29 (or score

    ≥20 without questions 15 to 21) at Beck Depression Inventory II (1996 version), the neuropsychologist doesn't conduct the battery of cognitive tests
14. Subject under curatorship or guardianship
15. Subject at which the initial cerebral MRI can't be achieved

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2012-06-29 (Actual); Study Completion 2016-07-26 (Actual)

PRIMARY OUTCOMES:
Demonstrate a significant improvement in HIV associated neurocognitive disorders after ARV intensification with increased CNS Penetration Effectiveness scoring ≥+3 and total CPE score ≥9. | Change from Baseline to Week 96
  HIV associated neurocognitive disorders classification with Frascati 3-stage

SECONDARY OUTCOMES:
Demonstrate a significant improvement in HIV associated neurocognitive disorders after ARV intensification with increased CNS Penetration Effectiveness scoring ≥+3 and total CPE score ≥9. | Change from Baseline to Week 48
  HIV associated neurocognitive disorders classification with Frascati 3-stage
To evaluate HIV associated neurocognitive disorders and Global Deficit Score change | Change from Baseline to Week 48
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification. Global Deficit Score (from 0 with no deficit to 5 with high neurocognitive disorder) is calculated with the results of 10 standardized battery tests.
To evaluate HIV associated neurocognitive disorders and Global Deficit Score change | Change from Baseline to Week 96
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification. Global Deficit Score (from 0 with no deficit to 5 with high neurocognitive disorder) is calculated with the results of 10 standardized battery tests.
To evaluate the evolution of HIV associated neurocognitive disorders with changes in CD4 and CD8 cells in plasma cells, and plasma HIV-1 viral loads | Change from Baseline to Week 48
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. CD4 and CD8 cells are measured in plasma with flow cytometry (results in cells/µL).
To evaluate the evolution of HIV associated neurocognitive disorders with changes in CD4 and CD8 cells in plasma cells, and plasma HIV-1 viral loads | Change from Baseline to Week 96
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. CD4 and CD8 cells are measured in plasma with flow cytometry (results in cells/µL).
To evaluate the evolution of HIV associated neurocognitive disorders with plasma HIV-1 viral load cells, and plasma HIV-1 viral loads | Change from Baseline to Week 48
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. Plasma HIV-1 viral load will be measured with an ultra-sensitive technique with a threshold of 5 copies/mL.
To evaluate the evolution of HIV associated neurocognitive disorders with plasma HIV-1 viral load cells, and plasma HIV-1 viral loads | Change from Baseline to Week 96
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. Plasma HIV-1 viral load will be measured with an ultra-sensitive technique with a threshold of 5 copies/mL.
To compare HIV associated neurocognitive disorders in HIV-1 infected patients with detectable and undetectable viral load in CSF | Day 0
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score.Detectable viral load in CSF is defined as a result >5 copies/mL with ultrasensitive HIV-RNA measure.
To compare HIV associated neurocognitive disorders in HIV-1 infected patients with detectable and undetectable viral load in CSF | Week 48
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score.Detectable viral load in CSF is defined as a result >5 copies/mL with ultrasensitive HIV-RNA measure.
To compare HIV associated neurocognitive disorders in HIV-1 infected patients with detectable and undetectable viral load in CSF | Week 96
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score.Detectable viral load in CSF is defined as a result >5 copies/mL with ultrasensitive HIV-RNA measure.
To evaluate the patterns of viral genotypic resistance in patients with virologic failure in blood or CSF | Week 12
  Virologic failure in the blood is defined as two results >100 copies/mL within one month. Virologic failure in the CSF is defined as a result >100 copies/mL
To evaluate the patterns of viral genotypic resistance in patients with virologic failure in blood or CSF | Week 24
  Virologic failure in the blood is defined as two results >100 copies/mL within one month. Virologic failure in the CSF is defined as a result >100 copies/mL
To evaluate the patterns of viral genotypic resistance in patients with virologic failure in blood or CSF | Week 36
  Virologic failure in the blood is defined as two results >100 copies/mL within one month. Virologic failure in the CSF is defined as a result >100 copies/mL
To evaluate the patterns of viral genotypic resistance in patients with virologic failure in blood or CSF | Week 48
  Virologic failure in the blood is defined as two results >100 copies/mL within one month. Virologic failure in the CSF is defined as a result >100 copies/mL
To evaluate the patterns of viral genotypic resistance in patients with virologic failure in blood or CSF | Week 60
  Virologic failure in the blood is defined as two results >100 copies/mL within one month. Virologic failure in the CSF is defined as a result >100 copies/mL
To evaluate the patterns of viral genotypic resistance in patients with virologic failure in blood or CSF | Week 72
  Virologic failure in the blood is defined as two results >100 copies/mL within one month. Virologic failure in the CSF is defined as a result >100 copies/mL
To evaluate the patterns of viral genotypic resistance in patients with virologic failure in blood or CSF | Week 84
  Virologic failure in the blood is defined as two results >100 copies/mL within one month. Virologic failure in the CSF is defined as a result >100 copies/mL
To evaluate the patterns of viral genotypic resistance in patients with virologic failure in blood or CSF | Week 96
  Virologic failure in the blood is defined as two results >100 copies/mL within one month. Virologic failure in the CSF is defined as a result >100 copies/mL
To evaluate the evolution of HIV associated neurocognitive disorders with the evolution of markers in CSF: neopterin, neurofilament light chain (NFL), CCL2, IL6, IL8, CXCL10, soluble CD14 | Change from Baseline to Week 48
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. CSF biomarkers were obtained using high-performance liquid chromatography coupled with fluorimetric detection for neopterin (nmol/L), using the Quanterix® single molecule array platform for neurofilament light protein (NF-L)(pg/mL), chemokine (C-C-motif) ligand-2 (CCL2)(pg/mL), interleukine 6 (IL6)(pg/mL), interleukine 8 (IL8)(pg/mL), chemokine (C-X-C-motif) ligand-10 (CXCL10)(pg/mL), and using an enzyme-linked immunosorbent assay (Biotechne®) for soluble CD14 (sCD14)(µg/mL) levels.
To evaluate the evolution of HIV associated neurocognitive disorders with the evolution of markers in CSF: neopterin, neurofilament light chain (NFL), CCL2, IL6, IL8, CXCL10, soluble CD14 | Change from Baseline to Week 96
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. CSF biomarkers were obtained using high-performance liquid chromatography coupled with fluorimetric detection for neopterin (nmol/L), using the Quanterix® single molecule array platform for neurofilament light protein (NF-L)(pg/mL), chemokine (C-C-motif) ligand-2 (CCL2)(pg/mL), interleukine 6 (IL6)(pg/mL), interleukine 8 (IL8)(pg/mL), chemokine (C-X-C-motif) ligand-10 (CXCL10)(pg/mL), and using an enzyme-linked immunosorbent assay (Biotechne®) for soluble CD14 (sCD14)(µg/mL) levels.
To evaluate the evolution of HIV associated neurocognitive disorders with the evolution of markers in plasma: neopterin, neurofilament light chain (NFL), CCL2, IL6, IL8, CXCL10, soluble CD14 | Change from Baseline to Week 48
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. Plasma biomarkers were obtained using high-performance liquid chromatography coupled with fluorimetric detection for neopterin (nmol/L), using the Quanterix® single molecule array platform for neurofilament light protein (NF-L)(pg/mL), chemokine (C-C-motif) ligand-2 (CCL2)(pg/mL), interleukine 6 (IL6)(pg/mL), interleukine 8 (IL8)(pg/mL), chemokine (C-X-C-motif) ligand-10 (CXCL10)(pg/mL), and using an enzyme-linked immunosorbent assay (Biotechne®) for soluble CD14 (sCD14)(µg/mL) levels.
To evaluate the evolution of HIV associated neurocognitive disorders with the evolution of markers in plasma: neopterin, neurofilament light chain (NFL), CCL2, IL6, IL8, CXCL10, soluble CD14 | Change from Baseline to Week 96
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. Plasma biomarkers were obtained using high-performance liquid chromatography coupled with fluorimetric detection for neopterin (nmol/L), using the Quanterix® single molecule array platform for neurofilament light protein (NF-L)(pg/mL), chemokine (C-C-motif) ligand-2 (CCL2)(pg/mL), interleukine 6 (IL6)(pg/mL), interleukine 8 (IL8)(pg/mL), chemokine (C-X-C-motif) ligand-10 (CXCL10)(pg/mL), and using an enzyme-linked immunosorbent assay (Biotechne®) for soluble CD14 (sCD14)(µg/mL) levels.
To evaluate HIV associated neurocognitive disorders and Brain MRI change | Change from Baseline to Week 48
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. Brain MRI is performed before and after ARV change
To evaluate HIV associated neurocognitive disorders and Brain MRI change | Change from Baseline to Week 96
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. Brain MRI is performed before and after ARV change
To compare sensitivity and specificity of the 2 screening tests (FAB test and Modified - HIV Dementia Scale) for the diagnosis of HAND | Day 0
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. Altered Frontal Assessment Battery test is defined with a score ≤15/18 and altered modified-HIV Dementia Scale screening test is defined with a score ≤10/12.
To evaluate regular monitoring of cognitive impairment by 10-items Cognitive Complaint Questionnaire to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 12
  10-items Cognitive Complaint Questionnaire is altered with a cutoff ≥3
To evaluate regular monitoring of cognitive impairment by 10-items Cognitive Complaint Questionnaire to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 24
  10-items Cognitive Complaint Questionnaire is altered with a cutoff ≥3
To evaluate regular monitoring of cognitive impairment by 10-items Cognitive Complaint Questionnaire to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 36
  10-items Cognitive Complaint Questionnaire is altered with a cutoff ≥3
To evaluate regular monitoring of cognitive impairment by 10-items Cognitive Complaint Questionnaire to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 48
  10-items Cognitive Complaint Questionnaire is altered with a cutoff ≥3
To evaluate regular monitoring of cognitive impairment by 10-items Cognitive Complaint Questionnaire to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 60
  10-items Cognitive Complaint Questionnaire is altered with a cutoff ≥3
To evaluate regular monitoring of cognitive impairment by 10-items Cognitive Complaint Questionnaire to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 72
  10-items Cognitive Complaint Questionnaire is altered with a cutoff ≥3
To evaluate regular monitoring of cognitive impairment by 10-items Cognitive Complaint Questionnaire to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 84
  10-items Cognitive Complaint Questionnaire is altered with a cutoff ≥3
To evaluate regular monitoring of cognitive impairment by 10-items Cognitive Complaint Questionnaire to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 96
  10-items Cognitive Complaint Questionnaire is altered with a cutoff ≥3
To evaluate regular monitoring of cognitive impairment by Inventory of Activity Daily Living part II to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 12
  Inventory of Activity Daily Living part II is altered with a cutoff ≥2
To evaluate regular monitoring of cognitive impairment by Inventory of Activity Daily Living part II to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 24
  Inventory of Activity Daily Living part II is altered with a cutoff ≥2
To evaluate regular monitoring of cognitive impairment by Inventory of Activity Daily Living part II to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 36
  Inventory of Activity Daily Living part II is altered with a cutoff ≥2
To evaluate regular monitoring of cognitive impairment by Inventory of Activity Daily Living part II to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 48
  Inventory of Activity Daily Living part II is altered with a cutoff ≥2
To evaluate regular monitoring of cognitive impairment by Inventory of Activity Daily Living part II to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 60
  Inventory of Activity Daily Living part II is altered with a cutoff ≥2
To evaluate regular monitoring of cognitive impairment by Inventory of Activity Daily Living part II to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 72
  Inventory of Activity Daily Living part II is altered with a cutoff ≥2
To evaluate regular monitoring of cognitive impairment by Inventory of Activity Daily Living part II to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 84
  Inventory of Activity Daily Living part II is altered with a cutoff ≥2
To evaluate regular monitoring of cognitive impairment by Inventory of Activity Daily Living part II to detect at the earliest possible changes in cognitive status | Change from Baseline to Week 96
  Inventory of Activity Daily Living part II is altered with a cutoff ≥2
To evaluate the Quality of Life during the study | Change from Baseline to Week 12
  Quality of Life is measured by Short Form 36 Health Survey
To evaluate the Quality of Life during the study | Change from Baseline to Week 24
  Quality of Life is measured by Short Form 36 Health Survey
To evaluate the Quality of Life during the study | Change from Baseline to Week 36
  Quality of Life is measured by Short Form 36 Health Survey
To evaluate the Quality of Life during the study | Change from Baseline to Week 48
  Quality of Life is measured by Short Form 36 Health Survey
To evaluate the Quality of Life during the study | Change from Baseline to Week 60
  Quality of Life is measured by Short Form 36 Health Survey
To evaluate the Quality of Life during the study | Change from Baseline to Week 72
  Quality of Life is measured by Short Form 36 Health Survey
To evaluate the Quality of Life during the study | Change from Baseline to Week 84
  Quality of Life is measured by Short Form 36 Health Survey
To evaluate the Quality of Life during the study | Change from Baseline to Week 96
  Quality of Life is measured by Short Form 36 Health Survey
To compare HIV associated neurocognitive disorders in patients with great CPE change ≥5 and patients with low CPE change (+3 or +4) | Change from Baseline to Week 48
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. CPE changes are analysed with most recent genotypic algorithm (v.2016)
To compare HIV associated neurocognitive disorders in patients with great CPE change ≥5 and patients with low CPE change (+3 or +4) | Change from Baseline to Week 96
  HIV associated neurocognitive disorders are measured with Frascati 3-stage classification and Global Deficit Score. CPE changes are analysed with most recent genotypic algorithm (v.2016)
To study the incidence and severity of adverse events during the study period | Week 12
  Neurologic or neuropsychologic adverse events are particularly analysed
To study the incidence and severity of adverse events during the study period | Week 24
  Neurologic or neuropsychologic adverse events are particularly analysed
To study the incidence and severity of adverse events during the study period | Week 36
  Neurologic or neuropsychologic adverse events are particularly analysed
To study the incidence and severity of adverse events during the study period | Week 48
  Neurologic or neuropsychologic adverse events are particularly analysed
To study the incidence and severity of adverse events during the study period | Week 60
  Neurologic or neuropsychologic adverse events are particularly analysed
To study the incidence and severity of adverse events during the study period | Week 72
  Neurologic or neuropsychologic adverse events are particularly analysed
To study the incidence and severity of adverse events during the study period | Week 84
  Neurologic or neuropsychologic adverse events are particularly analysed
To study the incidence and severity of adverse events during the study period | Week 96
  Neurologic or neuropsychologic adverse events are particularly analysed
To study the trough levels of antiretroviral drugs in blood and cerebrospinal fluid during the study | Day 0
  ARV concentrations were determined using an ultra-performance liquid chromatography coupled with tandem mass spectrometry
To study the trough levels of antiretroviral drugs in blood after ARV change | Week 4
  ARV concentrations were determined using an ultra-performance liquid chromatography coupled with tandem mass spectrometry
To study the trough levels of antiretroviral drugs in blood and cerebrospinal fluid during the study | Week 48
  ARV concentrations were determined using an ultra-performance liquid chromatography coupled with tandem mass spectrometry
To study the trough levels of antiretroviral drugs in blood and cerebrospinal fluid during the study | Week 96
  ARV concentrations were determined using an ultra-performance liquid chromatography coupled with tandem mass spectrometry
To study the cardiovascular risk evolution | Change from Baseline to Week 48
  Cardiovascular risk is measured with Framingham score, Systematic Coronary Risk Estimation, and D:A:D study model score
To study the cardiovascular risk evolution | Change from Baseline to Week 96
  Cardiovascular risk is measured with Framingham score, Systematic Coronary Risk Estimation, and D:A:D study model score are calcul

CONTACTS AND LOCATIONS:
Overall Officials: Philippe AEGERTER, Study Director — Clinical Research Unit
Locations (12):
- France (12):
  - Hôpital d'Argenteuil, Argenteuil
  - Hôpital Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier de Bligny, Briis-sous-Forges
  - Hôpital Mignot Centre Hospitalier de Versailles, Chesnay
  - Hôpital Raymond Poincaré, Garches
  - Centre Hospitalier de Gonesse, Gonesse
  - Institut Hospitalier Franco- Britannique, Levallois-Perret
  - Centre Hospitalier Marc Jacquet, Melun
  - Centre Hospitalier René Dubois, Pontoise
  - Hôpital Delafontaine, Saint-Denis
  - Centre Hospitalier Intercommunal de Poissy Germain en Laye, Saint-Germain-en-Laye
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No